CLINICAL TRIAL: NCT04823000
Title: Long Term Clinical and Immunological Effects of Repeated Mesenchymal Stem Cells (MSC) Injections in Patients With Progressive Forms of Multiple Sclerosis (MS)
Brief Title: Effects of Repeated Mesenchymal Stem Cells (MSC) in Patients With Progressive Multiple Sclerosis
Acronym: MSC-pMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-MS-001
Record Dates: First submitted 2021-01-11; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2020-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Mesenchymal Stem Cells
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Single Center, Open phase study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repeated MSCs treatment in MS patients (Experimental): Treatment with intrathecal and intravenous injection of autologous MSC (1 million cells per Kg of body weight)
  Interventions: Biological: Mesenchymal Stem Cells (MSC)

INTERVENTIONS:
Biological: Mesenchymal Stem Cells (MSC) — Repeated intrathecal and intravenous injection of autologous mesenchymal stem cells (1 million cells per Kg of body weight) at 6 months intervals.
  Other Names: MSC

SUMMARY:
An open prospective study with multiple (every 6-12 months) intrathecal or intravenous injections of autologous MSC in patients with progressive forms of MS (secondary progressive, primary progressive or relapsing-progressive), who failed to respond to first and second lines of immunomodulatory treatments and deteriorated (at least 0.5 degree in the EDSS scale) during the year preceding their inclusion to our study or had at least one major relapse without sufficient recovery.

DETAILED DESCRIPTION:
An open prospective study with multiple intrathecal or intravenous injections of autologous MSC in 24 patients with progressive forms of MS (secondary progressive, primary progressive or relapsing-progressive), who failed to respond to first and second lines of immunomodulatory treatments and deteriorated (at least 0.5 degree in the EDSS scale) during the year preceding their inclusion to our study or had at least one major relapse without sufficient recovery. Patients will be treated with 1x10 million MSC per kg of body weight, intrathecally and intravenously and subsequently with up to 8 courses of IT- or IV-injections of MSC (at the same dose), at intervals of 6-12 months. The duration of the trial is 4 years.

Patients will be followed up every 3 months for the whole duration of the trial, for safety assessment and changes in the disability scores (EDSS).

Immunological analysis will be performed at 4 time points (day 1, month 1, month 3 and month 6) following the first MSC-treatment and will include a fluorescent cell sorter (FACS) analysis to evaluate the proportions of the lymphocytes expressing markers of immune activation or of regulatory cell phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting patients fulfilling the Poser's criteria for definite MS
2. Age 18-70
3. Male and female
4. EDSS rate 5.5-7.5 (moderate to high disability)
5. Failure to two lines of the currently available registered immunomodulatory treatments for MS. The lack of response to these treatments was determined by either an increase in EDSS or the appearance of at least two relapses of MS during the year prior to inclusion.

Exclusion Criteria:

1. Patients who were treated with cytotoxic medications during the last three months prior to the infusion.
2. Patients suffering from significant cardiac, renal or hepatic failure or any other disease that may risk the patient or interfere with the ability to interpret the results.
3. Patients with active infections.
4. Patients with cognitive decline or inability to understand and sign the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Appearance of adverse events | 48 months following first treatment
  To evaluate the safety and tolerability of MSCs repeated treatment in progressive MS patients
The changes in Expanded Disability Status Scale (EDSS) score 0-10 scale, higher scores show worsening of disability) | 48 months
  To evaluate the changes in Expanded Disability Status Scale (EDSS) score after repeated MSC treatments compared to run-in period.

SECONDARY OUTCOMES:
Changes in the percentage of CD4/CD25/FoxP3 triple positive stained cells (T regulatory cells), following MSC-treatment | up to 6 months
  The percentage of CD4/CD25/FoxP3 triple positive stained cells, will be tested in the peripheral blood mononuclear cells obtained from MSC-treated patients using a fluorescent cell sorter (FACS) at 1 day, 1, 3 and 6 months post-MSC treatment and compared to baseline (before treatment) values for each patient. The mean post treatment values will be compared to the respective pre-treatmnent values at each time point.
Changes in the percentage of CD3+CD69+ cells (activated lymphocytes), following MSC-treatment | up to 6 months
  The percentage of CD3+CD69+ cells (activated lymphocytes), will be tested in the peripheral blood mononuclear cells obtained from MSC-treated patients using a fluorescent cell sorter (FACS) at 1 day, 1, 3 and 6 months post-MSC treatment and compared to baseline (before treatment) values for each patient. The mean post treatment values will be compared to the respective pre-treatmnent values at each time point.
Changes in the percentage of CD11c+/CD86+/Lin- cells (dendritic cells and antigen-presenting macrophages), following MSC-treatment | up to 6 months
  The percentage of CD11c+/CD86+/Lin- cells (dendritic cells and antigen-presenting macrophages), will be tested in the peripheral blood mononuclear cells obtained from MSC-treated patients using a fluorescent cell sorter (FACS) at 1 day, 1, 3 and 6 months post-MSC treatment and compared to baseline (before treatment) values for each patient. The mean post treatment values will be compared to the respective pre-treatmnent values at each time point.
Changes in the proliferation ability of mononuclear cells to PHA, following MSC-treatment | up to 6 months
  The proliferation ability of mononuclear cells to PHA will be tested in the peripheral blood mononuclear cells obtained from MSC-treated patients using a standard proliferative Thymidine-uptake assay at 1 day, 1, 3 and 6 months post-MSC treatment and compared to baseline (before treatment) values for each patient. The mean post treatment value (proliferation index) will be compared to the respective pre-treatmnent values at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Karussis, PhD, Principal Investigator — Hadassah HMO

REFERENCES:
- [Derived] Petrou P, Kassis I, Ginzberg A, Halimi M, Yaghmour N, Abramsky O, Karussis D. Long-Term Clinical and Immunological Effects of Repeated Mesenchymal Stem Cell Injections in Patients With Progressive Forms of Multiple Sclerosis. Front Neurol. 2021 May 31;12:639315. doi: 10.3389/fneur.2021.639315. eCollection 2021. PMID 34135843